CLINICAL TRIAL: NCT05348811
Title: Hepatic Arterial Infusion Chemotherapy (HAIC) Combined With Donafenib and Sintilimab in First-line Treatment of Unresectable Intrahepatic Cholangiocarcinoma (ICC): a Prospective, Open-label, Phase II Study
Brief Title: HAIC Combined With Donafenib and Sintilimab for Unresectable ICC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dean, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHANCE 2203
Record Dates: First submitted 2022-04-20; First posted 2022-04-27 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2022-06

CONDITIONS: Cholangiocarcinoma
Keywords: Hepatic arterial infusion chemotherapy; Donafenib; Sintilimab; Intrahepatic cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — donafenib; sintilimab

STUDY DESIGN:
Intervention Model Description: HAIC (GEMOX regimen) combined with donafenib and sintilimab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC combined with donafenib and sintilimab (Experimental): HAIC- GEMOX regimen, Day 1, every 3 weeks (Q3W). The maximum of 6 times.
  Sintilimab will be given on Day 1, 200 mg i.v. Q3W.The longest treatment time is 24 months.
  Donafenib was taken orally at 0.2 bid on an empty stomach, with an interval of about 12 hours. Donafenib treatment is initiated within 1 to 3 days of each HAIC treatment.
  Interventions: Drug: HAIC combined with donafenib and sintilimab

INTERVENTIONS:
Drug: HAIC combined with donafenib and sintilimab — HAIC- GEMOX regimen, gemcitabine 1000 mg/m2, oxaliplatin 85mg/m2 (if the maximum tumor diameter > 10cm, the dose is 130mg/m2), the first day of each cycle (D1), Q3W. The maximum of 6 times.
  Sintilimab will be given on the first day of each cycle (D1). 200 mg i.v. every 3 weeks until documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.The longest treatment time is 24 months.
  Donafenib was taken orally at 0.2 bid on an empty stomach (1 hour before or > 2 hours after meal) in the morning and evening of each administration day, with an interval of about 12 hours. Donafenib treatment is initiated within 1 to 3 days of each HAIC treatment until toxicity is intolerable, the investigator determines disease progression, death, informed consent is withdrawn, new antitumor therapy is initiated, or treatment is discontinued for any other reason specified in the protocol.
  Other Names: HAIC-donafenib-sintilimab

SUMMARY:
To evaluate the safety and tolerability of HAIC combined with donafenib and sintilimab in first-line treatment of unresectable ICC.

DETAILED DESCRIPTION:
Compared with systemic intravenous chemotherapy, hepatic arterial infusion chemotherapy(HAIC) has the advantages of improving local drug concentration and reducing toxic and side effects. Currently, it is gradually used in the treatment of intrahepatic cholangiocarcinoma (ICC) with good safety and high objective response rate. Immunotherapy combined with targeted and chemotherapy was well tolerated. At present, anti-programmed cell death protein-1(PD-1) antibody combined with chemotherapy and targeted therapy for advanced biliary tract tumors has initially shown good safety and encouraging efficacy, which is worthy of further exploration. Therefore, this study aims to evaluate the efficacy and safety of HAIC (GEMOX regimen) combined with donafenib and sintilimab in unresectable ICC.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic histologically or cytologically confirmed ICC
* No previous systemic treatment or local anti-tumor treatment other than surgery (biliary drainage is allowed), admission was allowed for more than 6 months after the end of adjuvant therapy
* Child-Pugh score ≤7
* Life expectancy ≥ 3 months
* At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST)1.1 criteria
* Eastern Cooperative Oncology Group(ECOG) performance status (PS) ≤ 1
* The functional indicators of important organs meet the following requirements:

  * Adequate blood count, liver-enzymes, and renal function: absolute neutrophil count ≥ 1.5*10^9 /L; platelet (PLT) ≥ 80 *10^9 /L; hemoglobin (HGB) ≥ 9.0 g/dL
  * Bilirubin ≤ 1.5 times upper limits of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 times ULN
  * Serum creatinine ≤ 1.5 times ULN, and creatinine clearance ≥ 60 ml/min (calculated by Cockcroft-Gault formula)
  * International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN
  * Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline of TSH is outside the normal range, patients with normal total T3 (or FT3) and free tetraiodothyronine (FT4) can also be enrolled
  * The myocardial enzyme profile was within the normal range
* For women who are not breastfeeding or pregnant, use contraception during treatment or 4 months after the end of treatment
* Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of the trial
* Patients who have signed Informed Consent Form (ICF) and are able to perform follow-up visits and the required procedures

Exclusion Criteria:

* Other malignancies diagnosed within 5 years before the first dose, excluding radically cured basal cell carcinoma of skin, squamous cell carcinoma of skin, and/or radically cured carcinoma in situ.
* Pathological diagnosis of hepatocellular carcinoma (HCC), mixed cholangiocarcinoma and HCC, and other malignant components of non-cholangiocarcinoma
* Receipt of treatment in other clinical trials within 4 weeks before the first dose
* Previous receipt of any antibody treatment involving anti-PD-1, anti-PD-L1/L2, or anti-CTLA4 or other immunotherapies
* Previous receipt of targeted drug(s)
* Previous receipt of palliative radiotherapy for biliary tract tumors, except for postoperative adjuvant radiotherapy
* Previous receipt of Chinese medicines with anti-tumor indications or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use to control pleural effusion) within 2 weeks before the first dose
* An active autoimmune disease requiring systemic therapy (e.g., palliative drugs, glucocorticoids, or immunosuppressants) developed within 2 years prior to first administration
* Have received systemic glucocorticoid therapy (excluding nasal spray, inhalation, or other topical glucocorticoid) or any other form of immunosuppressive therapy during the 4 weeks prior to the study
* Obstructive jaundice (active treatment, such as biliary drainage or stent, can be included after liver function recovery)
* Allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation is known
* Known allergic patients to sintilimab, the active ingredient of donafinib or excipients of the drug under study
* Not fully recovered from toxicity and/or complications associated with any intervention prior to initiation of treatment (i.e., ≤ grade 1 or baseline, excluding fatigue or hair loss)
* Human immunodeficiency virus (HIV), HIV 1/2 antibody positive
* Untreated active hepatitis B (defined as HBsAg positive with hepatitis B virus DNA (HBV-DNA) copy number greater than the ULN in the laboratory department of the research center) [Note: Hepatitis B patients who meet the following criteria can also be enrolled: 1) HBV DNA <2.5*10^3 copies/ml (500 IU/ml) before the first dose, should receive anti-HBV treatment throughout the study period; patients with anti-hepatitis B core antigen(HBc) (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), prophylactic anti-HBV therapy is not required, but viral reactivation needs to be closely monitored]
* Active HCV-infected subjects (HCV antibody positive and HCV-RNA level above the detection limit)
* Live attenuated vaccine was administered within 4 weeks prior to initial administration
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year)
* Presence of any serious or uncontrolled systemic disease, including but not limited to:

  * Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
  * Unstable angina pectoris, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) classification ≥ grade 2
  * Any arterial/venous thromboembolic events within 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient cerebral ischemic attack, pulmonary embolism, deep vein thrombosis, or any other history of serious thromboembolism
  * Receipt of major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks before the first dose or having unhealed wounds, ulcers, or fractures. Receipt of tissue biopsy or other minor surgeries within 7 days before the first dose, barring venipuncture and catheterization for intravenous infusion
  * Uncontrolled hypertension (systolic greater than 140 mmHg or diastolic greater than 90 mmHg) after optimal medical treatment, with the history of hypertensive crisis or hypertensive encephalopathy
  * Active tuberculosis
  * Active or poorly clinically controlled serious infections
  * Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction, gastrointestinal perforation, abdominal fistula within the past 6 months
  * Liver disease such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis
  * Poor control of diabetes (fasting blood glucose > 10 mmol/L)
  * Urine protein ≥ ++, and 24-hour urine protein quantification >1.0 g
  * With mental disorders and unable to cooperate with the treatment
* Unsuitable for enrollment judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | max 24 months
  According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for unresectable intrahepatic cholangiocarcinoma

SECONDARY OUTCOMES:
Disease control rate (DCR) | max 24 months
  The time from initiation of either regimen of combination therapy to all-cause death.
Duration of response (DOR) | max 24 months
  max 24 months
Progression-free survival (PFS) | max 24 months
  Time from initiation therapy to tumor progression according to the modified RECIST criteria or death from any cause.
Overall survival (OS) | max 42 months
  The time from initiation of either regimen of combination therapy to all-cause death.
Adverse events | max 42 months
  Adverse event (AE)、treatment emergent adverse event (TEAE)、serious adverse event (SAE).

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, Study Chair — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China